CLINICAL TRIAL: NCT02899598
Title: Genotyping of Human Platelet Alloantigens : Non-invasive Prenatal Diagnosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NEVER STARTED
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-55
Record Dates: First submitted 2016-09-09; First posted 2016-09-14 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Neonatal Thrombocytopenia Isoimmunization Maternal-fetal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pregnant women (Experimental)
  Interventions: Biological: Extra blood draw samples; Biological: extra amniotic fluid samples

INTERVENTIONS:
Biological: Extra blood draw samples — NEVER STARTED
Biological: extra amniotic fluid samples — NEVER STARTED

SUMMARY:
Neonatal thrombocytopenia isoimmunization maternal-fetal is related to maternal immunization against fetal platelet antigens with paternal origin not present in the mother. It is considered the equivalent of hemolytic disease of the newborn. The incidence of this disease is about 1 in 800-1000 births. The most severe forms associated petechiae, purpura or cephalhematoma at birth with a major risk of cerebral hemorrhages (20% to 25% of cases) can cause the death of the child (15%) or severe neurological troubles (15-30%) Biologic diagnosis requires the detection of anti-platelet antibodies with maternal determination of platelet phenotypes and genotypes of the two parents.

The objective of this work is to develop specific molecular tools to fetal platelet genotyping from maternal blood. We are particularly interested to antigens HPA-1, HPA-5 , HPA-3 and HPA-4. We evaluate the sensitivity and specificity of this test by comparing these results with those obtained from an invasive sampling of amniotic fluid.

This is a prospective study to assess the technical and diagnostic performance of a new molecular method noninvasive prenatal diagnosis of platelet genotyping.

DETAILED DESCRIPTION:
Neonatal thrombocytopenia isoimmunization maternal-fetal is related to maternal immunization against fetal platelet antigens with paternal origin not present in the mother. It is considered the equivalent of hemolytic disease of the newborn. The incidence of this disease is about 1 in 800-1000 births. The most severe forms associated petechiae, purpura or cephalhematoma at birth with a major risk of cerebral hemorrhages (20% to 25% of cases) can cause the death of the child (15%) or severe neurological troubles (15-30%) Biologic diagnosis requires the detection of anti-platelet antibodies with maternal determination of platelet phenotypes and genotypes of the two parents. When it is diagnosed, genetic counseling to the couple for a future pregnancy is necessary because the risk of recurrence is important and severity increases with the number of pregnancies. The risk depends on the nature of paternal antigens, homozygous or heterozygous. In case of heterozygosity, prenatal diagnosis is based on fetal platelet genotyping by an invasive procedure (amniocentesis or chorionic villus sampling) associated with a risk of fetal loss. The alloantibodies responsible for fetal damage are directed against platelet alloantigens: this is HPA system (human platelet alloantigen). 24 alloantigens have been described and 12 of them have a biallelic polymorphism (a: the most frequent allele and b the rare allele) divided into 6 groups (HPA-1, 2, 3, 4, 5, and 15). The genotype-phenotype correlations were performed for 22 of the 24 alloantigens and show that the antigenic polymorphism results from the presence of a SNP (single nucleotide polymorphism-).

In 1997, Lo et al showed the presence of 3-6% of fetal DNA in maternal blood. This discovery led to the development of methods of non-invasive prenatal diagnosis: 1/ the determination of fetal Rhesus 2/ fetal sex by real-time quantitative PCR.

The objective of this work is to develop specific molecular tools to fetal platelet genotyping from maternal blood. We are particularly interested to antigens HPA-1, HPA-5 , HPA-3 and HPA-4. We evaluate the sensitivity and specificity of this test by comparing these results with those obtained from an invasive sampling of amniotic fluid.

This is a prospective study to assess the technical and diagnostic performance of a new molecular method noninvasive prenatal diagnosis of platelet genotyping.

ELIGIBILITY:
Inclusion Criteria:

* patients with known risk of platelet alloimmunization
* patients for whom suspicion of fetal cerebral hemorrhage has been advanced on ultrasound or fetal MRI signs

Exclusion Criteria:

* Twin pregnancy or triple

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-27 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
number of Fetomaternal platelet incompatibilities detected | 30 months

CONTACTS AND LOCATIONS:
Overall Officials: Urielle Desalbres, Study Director — Assistance Publique Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No